CLINICAL TRIAL: NCT01061957
Title: Clinical, Virological and Immunological Course in Danish Patients With Triple Class Failure Receiving Raltegravir as Part of a Salvage Regimen.
Brief Title: Raltegravir Treatment in Patients Failing Highly Active Antiretroviral Therapy (HAART) in Denmark
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Jan Gerstoft, MD, Professor, The Danish HIV Cohort Study
Other Study IDs: 37593
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-01

CONDITIONS: HIV Infections
Keywords: Treatment outcome; HIV treatment
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Raltegravir patients: HIV patients who initiated raltegravir due to virological failure
- Haart naive patients: HIV patients initiating HAART for the first time

SUMMARY:
Raltegravir is the first integrase inhibitor approved for treatment of HIV infected patients harboring multiresistant viruses. The drug has been proved effective in both trials and clinical settings, but the long-term efficacy is not described and the effect compared to treatment in Highly active antiretroviral therapy (HAART) naive patients remains to be established.

DETAILED DESCRIPTION:
Highly active antiretroviral therapy (HAART) was introduced more than a decade ago and the therapy has decreased mortality and morbidity of HIV patients dramatically. The first HAART regimens were combined of nucleoside reverse transcriptase inhibitors (NRTIs), non-nucleoside reverse transcriptase inhibitors (NNRTIs) and protease inhibitors (PIs). Especially the early regimes carried a substantial risk of failure and subsequent development of resistance to the three drug classes. Thus there has been a need for development of new drugs with activity against viruses resistant to the classical HAART regimens either as new drugs from the old classes without (or with limited) cross resistance to the older compounds or drugs from new classes with new antiretroviral mechanisms. The optimal choice for salvage therapy for HIV infected patients has been shown to require at least two, and preferably three, fully active drugs. Until recently, salvage regimens used to treat patients harbouring multidrug-resistant HIV generally included only one new agent from the classic drug classes added to an optimized background therapy which did not contain any fully active agents. This approach, conditioned by limited drug options, put patients at high risk of virological failure and resistance to the new agent, as well as to other agents in the same drug classes. A breakthrough has been the resent development of integrase inhibitors, which is a new class of antiretroviral drugs. One of these drugs - raltegravir - has demonstrated its activity in patients with virological failure on classical antiretroviral drugs. In the BENCHMARK randomized clinical trials, which were conducted in HIV-infected patients with limited treatment options, 62% of patients taking raltegravir plus optimized background treatment achieved plasma HIV RNA levels <50 copies/mL at week 48. Although the drug - often used together with other new drugs - has been proved effective in clinical trials and recently in "real life" clinical settings, the long-term efficacy is not described and the effect compared to treatment in HAART naive patients remains to be established. In a nationwide cohort of HIV infected patients, we identified the patients, who initiated raltegravir due to virological failure and a matched control cohort of patients initiating HAART for the first time. We compared these two cohorts with respect to virological suppression, gain in CD4 count and time to first change of initial regimen.

ELIGIBILITY:
Inclusion Criteria:

* Raltegravir cohort patients: From the Danish HIV Cohort Study (DHCS) we included all HIV-1 positive patients, who

  1. started raltegravir after 1 January 2006 and before 1 July 2009,
  2. had been treated with HAART previously
  3. had at least two VL tests done prior to initiation of raltegravir treatment,
  4. had virological failure prior to start of raltegravir and
  5. did not participate in randomized clinical trials on raltegravir. Virological failure was defined as VL > 500 copies/ml in the two latest VL tests prior to raltegravir initiation while on HAART treatment.
* Control cohort patients: From DHCS we identified a control cohort of HIV infected patients who started HAART for the first time after 1 January 2006 and before 1 July 2009. From this population we extracted two control patients for each raltegravir patient, each matched by gender, race (Caucasian, Black and other), route of HIV infection (homosexual, heterosexual, injection drug user (IDU) and other) and age (intervals of < 20 years, 20 to 30 years, 30 to 40 years, > 50 years).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: One cohort of HIV patients with virological failure initiating Raltegravir One control cohort of HIV patients initiating HAART for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2006-01; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
virological suppression and CD4 cell gain | 3,5 years

SECONDARY OUTCOMES:
Time to first change of initial regimen. | 3,5 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Danish HIV Cohort Study, Rigshospitalet, Copenhagen, Denmark